CLINICAL TRIAL: NCT04426149
Title: Clinical Effects of Oral Trehalose In Patients With Spinocerebellar Ataxia 3: A Pilot Study
Brief Title: Clinical Effects of Oral Trehalose In Patients With Spinocerebellar Ataxia 3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Malaysia (Other)
Responsible Party: Principal Investigator, Dr Norlinah Mohamed Ibrahim, Professor, National University of Malaysia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UKM PPI/111/8/JEP-2017-826
Record Dates: First submitted 2019-04-18; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Spinocerebellar Ataxia 3
MeSH Terms: conditions — Machado-Joseph Disease | interventions — Trehalose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- interventional (Experimental): supplement: trehalose
  Interventions: Dietary Supplement: trehalose

INTERVENTIONS:
Dietary Supplement: trehalose — patients were instructed to ingest 100g of oral trehalose diluted in 500ml of water or other beverages daily

SUMMARY:
There are no clinically established treatments which have been proven to delay the disease progression in spinocerebellar ataxia (SCA) 3. Most available treatments are only for symptom alleviation, and thus the majority of patients will eventually progress to needing and wheel chair and eventually bedridden.

As trehalose appear to be potentially promising treatment in SCA, the investigators aim to conduct this study using oral trehalose in our genetically confirmed SCA 3 patients.

DETAILED DESCRIPTION:
This prospective single arm interventional study involved 13 genetically confirmed spinocerebellar ataxia (SCA) 3 patients with no concomitant diabetes, over 6 months. Following baseline assessment, patients were instructed to ingest 100g of oral trehalose diluted in 500ml of water or other beverages daily. Assessments were performed at baseline, 2, 4 and 6 months using ataxia rating scales (SARA, SCAFI and INAS) and EQ-5D-3L scale for quality of life assessment.

ELIGIBILITY:
Inclusion Criteria:

1. DNA diagnosis of SCA 3 in the study subject of his/ her affected family member(s)
2. Consent to participate in the study
3. The age of 18 years and older

Exclusion Criteria:

1. Unconfirmed SCA 3
2. Concomitant disorder(s) that affect SARA and other ataxia measures used in this study
3. Diabetes
4. Malabsorption of trehalose underlies intolerance to mushrooms, since the lack of absorption results in diarrhoea and intestinal distress.
5. Less than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2018-09-07 (Actual); Study Completion 2018-09-07 (Actual)

PRIMARY OUTCOMES:
scale of rating of ataxia (SARA) score months, | 2 monthly intervals for 6 months
  Assessment of SARA scores by a single assessor
SCA Functional Index Scores | 2 monthly intervals for 6 months
  Assessment of SCAFI by a single assessor
EQ5D3L - quality of life scores | 2 monthly intervals for 6 months
  Assessment of quality of life scores

SECONDARY OUTCOMES:
Side effects Profile | 2 monthly intervals for 6 months
  Adverse Effects
Blood investigation | At baseline and at 6 months
  Measurement of renal profile, fasting blood glucose, full blood count and liver profile

CONTACTS AND LOCATIONS:
Overall Officials: NORLINAH MOHAMED IBRAHIM, MBBCH, Principal Investigator — norlinah@ppukm.ukm.edu.my
Locations (1):
- Pusat Perubatan Universiti Kebangsaan Malaysia, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No